CLINICAL TRIAL: NCT06306950
Title: Optimization of Cerebral Oximetry And Avoid Cerebral Deoxygenation In Severe Traumatic Brain Injury.
Brief Title: Prioritization of Cerebral Deoxygenation in Severe Traumatic Brain Injury and Mortality Benefit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PMK-00098
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Hypoxia; Severe Traumatic Brain Injury
Keywords: Severe Traumatic Brain Injury; Cerebral Desaturation; Regional Cerebral Oxygen Saturation; Neurosurgical Intensive Care Unit
MeSH Terms: conditions — Hypoxia, Brain; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: In a prospective study, 80 patients were randomized to either application of near-infrared reflectance spectroscopy (NIRS) monitoring with active display or attempt to make an intervention to keep regional cortical cerebral oxygen saturation (rSO2) ≥ 55% by increased cardiac output, mean arterial pressure, and adjusting the ventilator to hypoventilation (PaCO2 40-45 mmHg) (exclude in radiographic brain herniation) (intervention, n = 40), compared with usual care (n = 40). Clinical outcomes were assessed by a blind observer. Data collection comprised of patients' demographic data, intervention process, and outcomes of treatment assessed by modified Rankin scale (mRS) followed up at 1 year.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Upon arrival in the emergency department, the randomization envelope was opened, and patients were assigned into either active treatment (intervention) or usual care (control) groups with cerebral oximetry monitoring using NIRS bilaterally (Root; Prime Medical Corporation, MASIMO, USA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near infrared spectroscopy neuromonitor (Experimental): Patients were assigned into active treatment (intervention) with cerebral oximetry monitoring using Near infrared spectroscopy monitoring (NIRS) bilaterally (Root; Prime Medical Corporation, MASIMO, USA). After cleansing the adjacent skin area with alcohol, an adhesive optode pad was placed over each frontal to temporal area. Resting baseline rSO2 values were obtained after waiting at least 1 minute after the placement of the sensors. Once values had stabilized, the screen was electronically blinded, and the time monitoring and baseline parameters were recorded by taking the data frequency of 1 minute, 3 minutes after the start recording. For the intervention group, an alarm threshold at 55% of the resting baseline rSO2 value was established. Continuous rSO2 values were stored on a floppy disk with a 15-second update for the duration of the perioperative period.
  Interventions: Device: Near infrared spectroscopy neuromonitor to prevent cerebral desaturation
- No neuromonitor (No Intervention): For usual care patients, the best clinical practices aim at maintaining hemoglobin (Hb) levels greater than 7 g/dl, blood glucose within the institutional normal range of 80-180 mg/dl, and mean arterial pressure (MAP) of 65 mmHg in the ICU and were monitored for invasive arterial blood pressure, peripheral O2 saturation (SpO2), and electrocardiograms. Sedative and paralysis agents were given; keep the Richmond Agitation Sedation Scale (RASS) less than -3 and the Bispectral Index (BIS) 40-60 monitoring based on bedside intensivist judgment, including fentanyl, propofol, midazolam, and cisatracurium. Patients were mechanically ventilated using a volume-control ventilation mode with a tidal volume of 8 ml/kg, a respiratory rate adjusted to maintain normocapnia, an inspired oxygen fraction adjusted to maintain SpO2 above 95%, and an inspiratory/expiratory ratio of 1:2.

INTERVENTIONS:
Device: Near infrared spectroscopy neuromonitor to prevent cerebral desaturation — patients were assigned into active treatment (intervention) or usual care (control) groups with cerebral oximetry monitoring using NIRS bilaterally (Root; Prime Medical Corporation, MASIMO, USA) [17]. After cleansing the adjacent skin area with alcohol, an adhesive optode pad was placed over each frontal to temporal area. Resting baseline rSO2 values were obtained after waiting at least 1 minute after the placement of the sensors.
  Arms: Near infrared spectroscopy neuromonitor

SUMMARY:
Severe traumatic brain injury with a decrease in cerebral oximetry is associated with multiple impaired systemic microcirculations, more morbidities, and a higher mortality rate. When using the brain as an index organ, interventions to improve brain oxygen delivery may have systemic benefits for these patients.

DETAILED DESCRIPTION:
We conducted a prospective interventional study. Data from all 80 severe traumatic brain injury patients were randomized to either perioperative cerebral regional oxygen saturation (rSO2) monitoring with an intervention protocol to prevent cerebral desaturation (intervention, n = 40), or underwent blinded rSO2 monitoring (control, n = 40). Predefined clinical outcomes were assessed by a blinded observer. 40 were retrieved on April 1, 2021 to February 28, 2024. Data collection comprised of patients' demographic data, treatment process, and outcomes of treatment was implemented in the intensive care unit. The pre-intervention included all consecutive severe traumatic brain injury patients admitted as participants. After ethic approval in all methods and obtaining written informed consent from the legal relatives, severe traumatic brain injury patients were enrolled on the basis of inclusion criteria of age ≥ 20 years, Patients were recruited from the preoperative clinic in cases of neurosurgery with agreement. Upon arrival in the emergency department, the randomization envelope was opened, and patients were assigned into either active treatment (intervention) or usual care (control) groups with cerebral oximetry monitoring using NIRS bilaterally (Root; Prime Medical Corporation, MASIMO, USA). After cleansing the adjacent skin area with alcohol, an adhesive optode pad was placed over each frontal to temporal area. Resting baseline rSO2 values were obtained after waiting at least 1 minute after the placement of the sensors. Once values had stabilized, the screen was electronically blinded, and the time monitoring and baseline parameters were recorded by taking the data frequency of 1 minute, 3 minutes after the start recording. For the intervention group, an alarm threshold at 55% of the resting baseline rSO2 value was established. Continuous rSO2 values were stored on a floppy disk with a 15-second update for the duration of the perioperative period. With the application of the scalp dressing and before leaving the ICU, monitoring was discontinued, and optodes were removed after discharge from the ICU for 10 days.

For all severe traumatic brain injury patients, the best clinical practices aim at maintaining hemoglobin (Hb) levels greater than 7 g/dl, blood glucose within the institutional normal range of 80-180 mg/dl, and mean arterial pressure (MAP) of 65 mmHg in the intensive care unit. In the intervention group, a prioritized management protocol was used to maintain rSO2 values at or above 55% of the baseline threshold. With a decrease in rSO2, the patient's head position was checked to ensure that it had not been rotated or kinked, and the face was observed to detect plethora. If PaCO2 or end-tidal CO2 was below 40 mmHg during positive pressure ventilation, ventilation was reduced to achieve PaCO2 ≥ 40 mmHg. If MAP was < 65 mmHg, 40 μg increments of intravenous norepinephrine were administered to achieve an MAP ≥ 65 mmHg. If the cardiac index was < 2.0 L/m2/min, administration of dobutamine increased to 2.5 L/m2/min. In patients with persistent rSO2 below the treatment threshold, FiO2 was increased. If Hb was below 7 g/dl, a red blood cell transfusion was administered immediately. Cerebral oximetry monitoring was continued after discharge from the intensive care unit for 10 days. To maintain participant blindness, no study group identifiers were included with the patient or in the patients' charts. For neurosurgical intensive care unit postoperatively, all patients were transferred to an autonomous, protocol-given, "closed" neuro-intensive care unit under the exclusion care of an intensive care unit intensivist without direct reference to the attending neurosurgeons or anesthesiologists. Criteria for discharge from the intensive care unit comprised (1) hemodynamic stability defined as absence of vasopressor or inotropic drugs, removal of arterial and pulmonary artery or central venous catheters, and absence of cardiac arrhythmias; (2) post-extubation respiratory parameter adequacy with maintenance of pulse oximetry (SpO2) > 95% with supplemental O2 below 5 L/min; (3) level of consciousness appropriate sufficient to protect their airway; and (4) good kidney function (urinary output ≥ 0.5 mL/kg/hr). Data on ICU admission and discharge times, and use of a vasopressor were obtained from the intensive care unit database.

The sample size was based upon a projected near infrared spectroscopy (NIRS)-derived tissue oxygenation published in Annual Intensive Care 2012 about the correlation between near infrared spectroscopy (NIRS) in anesthesia and intensive care and brain tissue oxygenation and major organ function. As a priority assumption, we hypothesized that a 50% reduction in the incidence of overall complications would be associated with active NIRS cerebral oximetry. Accepting a p-value < 0.05 for statistical significance and a β error of 0.2, we determined that 40 patients in each group were required for this study. The randomization method was done by blinded envelopes assigning treatment allocation and placing them in computer-generated random order, which were written in order to sequentially identify each subject that registered in this protocol and was disclosed in the neurosurgical ICU. Cerebral deoxygenation means a reduction in saturation below 55% of baseline for 1 minute or longer. To minimize the probability of patients reaching these levels, interventions to improve cerebral oxygenation were administered when rSO2 decreased to < 55% of baseline for > 15 s. Mean and minimum values of rSO2. Categorical values are presented as numbers (percentage) and were analyzed using contingency table analysis, Fisher's exact test, χ2, and Wilcoxon's rank sum tests as appropriate. Continuous variables are presented as mean ± SD using an unpaired t-test or ANOVA for analysis, with a p-value < 0.05 required for statistical significance.

80 patients in the ICU were monitored for invasive arterial blood pressure, peripheral O2 saturation (SpO2), and electrocardiograms. Sedative and paralysis agents were given; keep the Richmond Agitation Sedation Scale (RASS) less than -3 and the Bispectral Index (BIS) 40-60 monitoring based on bedside intensivist judgment, including fentanyl, propofol, midazolam, and cisatracurium. Patients were mechanically ventilated using a volume-control ventilation mode with a tidal volume of 8 ml/kg, a respiratory rate adjusted to maintain normocapnia, an inspired oxygen fraction adjusted to maintain SpO2 above 95%, and an inspiratory/expiratory ratio of 1:2. The inclusion criteria were age more than 20 years old, Severe traumatic brain injury defined as Glasgow coma scale < 8, and the exclusion criteria were patients who had a pregnancy, an infection at the forehead, a status epilepticus, a history of drug addiction, and Severe traumatic brain injury combination with metabolic causes.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years old
* severe traumatic brain injury defined as Glasgow coma scale < 8

Exclusion Criteria:

* pregnancy
* infection at the forehead
* status epilepticus
* history of drug addiction
* severe traumatic brain injury combination with metabolic causes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) followed up at 1 year | 1 year
  Documentation in the medical record of a Modified Rankin Score (mRS). The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.

CONTACTS AND LOCATIONS:
Overall Officials: PANU BOONTOTERM, MD., FRCNST, Principal Investigator — Phramongkutklao College of Medicine and Hospital; Suthee Panichkul, MD., Study Director — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao College of Medicine and Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The data sets used and/or analysed during the current study are available from the corresponding author on reasonable request. The data are not publicly available due to information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Roldan M, Kyriacou PA. Near-Infrared Spectroscopy (NIRS) in Traumatic Brain Injury (TBI). Sensors (Basel). 2021 Feb 24;21(5):1586. doi: 10.3390/s21051586. PMID 33668311
- [Result] Davies DJ, Su Z, Clancy MT, Lucas SJ, Dehghani H, Logan A, Belli A. Near-Infrared Spectroscopy in the Monitoring of Adult Traumatic Brain Injury: A Review. J Neurotrauma. 2015 Jul 1;32(13):933-41. doi: 10.1089/neu.2014.3748. Epub 2015 Apr 17. PMID 25603012
- [Result] Sen AN, Gopinath SP, Robertson CS. Clinical application of near-infrared spectroscopy in patients with traumatic brain injury: a review of the progress of the field. Neurophotonics. 2016 Jul;3(3):031409. doi: 10.1117/1.NPh.3.3.031409. Epub 2016 Apr 25. PMID 27226973
- [Result] Viderman D, Ayapbergenov A, Abilman N, Abdildin YG. Near-infrared spectroscopy for intracranial hemorrhage detection in traumatic brain injury patients: A systematic review. Am J Emerg Med. 2021 Dec;50:758-764. doi: 10.1016/j.ajem.2021.09.070. Epub 2021 Oct 3. PMID 34879500
- [Result] Mathieu F, Khellaf A, Ku JC, Donnelly J, Thelin EP, Zeiler FA. Continuous Near-infrared Spectroscopy Monitoring in Adult Traumatic Brain Injury: A Systematic Review. J Neurosurg Anesthesiol. 2020 Oct;32(4):288-299. doi: 10.1097/ANA.0000000000000620. PMID 31306264
- [Result] Fawaz R, Laitselart P, Morvan JB, Riff JC, Delmas JM, Dagain A, Joubert C. Application of near-infrared spectroscopy to triage of traumatic brain injuries in high-intensity conflicts. BMJ Mil Health. 2024 May 22;170(3):273-274. doi: 10.1136/military-2022-002301. No abstract available. PMID 36600643
- [Result] Brogan RJ, Kontojannis V, Garara B, Marcus HJ, Wilson MH. Near-infrared spectroscopy (NIRS) to detect traumatic intracranial haematoma: A systematic review and meta-analysis. Brain Inj. 2017;31(5):581-588. doi: 10.1080/02699052.2017.1287956. Epub 2017 Apr 25. PMID 28440675